CLINICAL TRIAL: NCT01602926
Title: Randomized Prospective Trial of Minimally Invasive Surgery Versus Standard Surgery for Correction of Hallux Valgus.
Brief Title: Prospective Trial of Minimally Invasive Surgery Versus Standard Surgery for Correction of Hallux Valgus
Acronym: Minibunion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henry DeGroot, M.D. (Other)
Responsible Party: Principal Investigator, Henry DeGroot, P.I., Henry DeGroot, M.D.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2012-Minibunion
Record Dates: First submitted 2012-05-15; First posted 2012-05-21 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Hallux Valgus
Keywords: hallux valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional surgery arm (Experimental): The conventional surgical technique is a Chevron-type distal metatarsal osteotomy, which is performed through a dorsomedial incision approximately 7 cm long. And osteotomy of the distal portion of the first metatarsal is made. The capital or distal fragment of the metatarsal is mobilized and displaced laterally an adequate amount to correct the hallux valgus deformity. The capital or distal fragment is stabilized in corrected position with screws.
  Interventions: Procedure: conventional surgical technique - Chevron-type distal metatarsal osteotomy
- minimally invasive technique (Experimental): The minimally invasive surgical technique is a transverse subcapital distal metatarsal osteotomy, which is performed through a direct medial incision approximately 1 cm long. The osteotomy of the distal portion of the first metatarsal is made using fluoroscopic image guidance. The capital or distal fragment of the metatarsal is mobilized and displaced laterally an adequate amount to correct the hallux valgus deformity. A 2.0 mm Kirschner wire is placed percutaneously in a position medial to the proximal phalanx, and advanced proximally using fluoroscopic guidance until the proximal end of the wire is located in a stable position within the medullary cavity of the first metatarsal
  Interventions: Procedure: minimally invasive surgical technique

INTERVENTIONS:
Procedure: conventional surgical technique - Chevron-type distal metatarsal osteotomy — The conventional surgical technique is a Chevron-type distal metatarsal osteotomy, which is performed through a dorsomedial incision approximately 7 cm long. And osteotomy of the distal portion of the first metatarsal is made. The capital or distal fragment of the metatarsal is mobilized and displaced laterally an adequate amount to correct the hallux valgus deformity. The capital or distal fragment is stabilized in corrected position with screws. The internal fixation screws used in the conventional surgical technique do not require removal.
  Arms: conventional surgery arm
Procedure: minimally invasive surgical technique — The minimally invasive surgical technique is a transverse subcapital distal metatarsal osteotomy, which is performed through a direct medial incision approximately 1 cm long. The osteotomy of the distal portion of the first metatarsal is made using fluoroscopic image guidance. The capital or distal fragment of the metatarsal is mobilized and displaced laterally an adequate amount to correct the hallux valgus deformity. A 2.0 mm Kirschner wire is placed percutaneously in a position medial to the proximal phalanx, and advanced proximally using fluoroscopic guidance until the proximal end of the wire is located in a stable position within the medullary cavity of the first metatarsal (see figures) .The distal end of the Kirschner wire is left outside the skin where it is cut to length and covered. The Kirschner wire is removed after six weeks.
  Arms: minimally invasive technique
Procedure: minimally invasive surgical technique — The minimally invasive surgical technique is a transverse subcapital distal metatarsal osteotomy, which is performed through a direct medial incision approximately 1 cm long. The osteotomy of the distal portion of the first metatarsal is made using fluoroscopic image guidance. The capital or distal fragment of the metatarsal is mobilized and displaced laterally an adequate amount to correct the hallux valgus deformity.
  Arms: minimally invasive technique

SUMMARY:
Hallux valgus is a common deformity of the big toe, defined as medial deviation of the first metatarsal bone along with lateral deviation of the first toe. Surgery has been shown to be beneficial when compared to orthotics or no treatment. While generally effective, surgery is associated with significant post-operative pain and disability, with several weeks of limited mobility. Minimally invasive techniques have the potential to lead to increased patient satisfaction while still achieving adequate correction of the deformity.

This trial is a non-inferiority treatment study, with open-label, randomized, prospective, controlled, parallel experimental design, to compare the clinical and radiographic outcomes of a minimally invasive surgery versus a conventional surgery for hallux valgus. This trial examines two different surgical interventions. No drug or device is being evaluated in this trial.

60 to 100 patients, over the age of 18 years, undergoing surgical correction of mild to moderate hallux valgus will be enrolled in the trial. The patients will be randomized to two groups, one treated with a conventional distal osteotomy surgery, the other treated with a minimally invasive surgery. Randomization will occur immediately prior to surgery via a multitude of opaque envelopes containing a coded group assignment. Due to the differences in the techniques, neither the investigator and the subject can be effectively blinded to the group assignment. Data collection for the outcomes measures will occur preop, and then post of at 2 weeks, 12 weeks, and at 1,2, and 3 years.

The primary outcomes measure is the Manchester-Oxford Foot Questionnaire Score (MOXFQ). Manchester-Oxford Foot Questionnaire' (MOXFQ), a 16 item patient-reported questionnaire consisting of three domains/scales: 'Walking/standing' (seven items), 'Pain' (five items) and 'Social interaction' (four items). The MOXFQ is a validated disease-specific outcomes scale for foot and ankle surgery which has been shown to be responsive and reliable.

Secondary outcome measures are preoperative to postoperative change in hallux valgus angle (HVA). Radiographic outcomes parameters will be measured using weight-bearing radiographs to analyze preoperative and postoperative hallux valgus angle, and the correction or normalization thereof. (Degrees of correction = 2 week preoperative HVA - 12 week postoperative HVA.)

DETAILED DESCRIPTION:
Randomized prospective trial of minimally invasive surgery versus standard surgery for correction of hallux valgus.

Introduction

It is estimated that more than 200,000 hallux valgus surgeries are performed each year in the United States. [1] More than 100 procedures have been described for correction of hallux valgus.[2] Considerable controversy remains over the best technique.

Recently, a number of minimally invasive techniques for correction of hallux valgus have been described. [3, 5, 6]. These minimally invasive techniques emphasize less traumatic surgical exposure and more limited dissection of the soft tissues. It has been proposed that minimally invasive procedures lead to less pain, decreased swelling, shorter recovery times and more rapid return to full weightbearing activities. Not all reports have been positive, and some authors report an increased number of complications, including loss of correction and malposition of the bones [7].

Minimally invasive treatment of hallux valgus is becoming increasingly common in podiatric and orthopedic clinical practice, due to the theoretical advantages of more rapid recovery, more rapid return to full activities, and decreased pain. These techniques have the potential advantage of providing better clinical outcomes and having lower cost.

An increasing number of research publications on this topic have appeared in recent years, which reflects both growing interest and development in this field amongst foot and ankle surgeons. However, despite the increasing interest, there are no high-quality studies of these procedures available. In a 2011 systematic review [8], 24 publications describing the outcomes of minimally invasive hallux valgus surgery were identified and analyzed. All the studies were level IV quality (case series, with the exception of two that were level III (a retrospective comparative studies). No randomized prospective controlled studies have been published, and validated disease-specific outcomes measures are seldom used [9].

No high quality trials of any minimally invasive techniques have been published, and as a result, basic questions still remain unanswered: Do minimally invasive procedures have fewer complications than standard procedures? Are minimally invasive procedures associated with superior patient-based outcomes? Are the radiographic outcomes of minimally invasive techniques equivalent? Randomized, prospective clinical trials are required, utilizing validated outcomes measures.

Study Objectives

To compare the patient-based outcomes and radiographic outcomes of minimally invasive surgery versus standard surgery for correction of hallux valgus.

Primary Outcomes Measure

The primary outcomes measure is the Manchester-Oxford Foot Questionnaire Score (MOXFQ). Manchester-Oxford Foot Questionnaire' (MOXFQ), a 16 item patient-reported questionnaire consisting of three domains/scales: 'Walking/standing' (seven items), 'Pain' (five items) and 'Social interaction' (four items). The MOXFQ is a validated disease-specific outcomes scale for foot and ankle surgery which has been shown to be responsive and reliable. In observational studies, minimal clinically important difference (MCID) for the various domains of the MOXFQ were 16, 12, and 24 for the MOXFQ Walking/standing, Pain, and Social Interaction domains, respectively. The MOXFQ has demonstrated good responsiveness when compared with the AOFAS forefoot score. Statistical analysis of the data will show if the null hypothesis that there are no statistically significant differences between groups with respect to the postoperative MOXFQ scores at 12 weeks, 1 year, 2 years and 3 years is rejected.

Secondary outcome measures are preoperative to postoperative change in hallux valgus angle (HVA). Radiographic outcomes parameters will be measured using weight-bearing radiographs to analyze preoperative and postoperative hallux valgus angle, and the correction or normalization thereof. (Degrees of correction = preoperative HVA - 12 week postoperative HVA.)

Statistical analysis of the data will show if the null hypothesis that there are will be no statistically significant differences between groups with respect to the degree of correction of the hallux valgus angle is rejected.

Study Design

Type

Non-inferiority treatment study, open-label, randomized, prospective, controlled, parallel experimental design.

Location

Study-related patient visits will take place in the office of the principal investigator, Dr. Henry DeGroot, white 544, Newton Wellesley Hospital MOB Surgery will take place in the operating rooms at the Newton Wellesley Hospital. Post operative evaluations will take place in the office of the principal investigator and in the Newton Wellesley Hospital cast room. Preoperative and postoperative x-rays will take place in the radiology department of the Newton Wellesley Hospital.

Duration

Subjects will be enrolled until sufficient numbers have been achieved for the two groups, which is estimated to require 36 months. The time of active participation for each subject will be 12 weeks.

The period of long-term follow-up for each subject will be 36 months, beginning from the date of surgery.

Research Plan

Study Intervention

The study will compare two surgical techniques for correction of hallux valgus, which are detailed below. Other than the intraoperative surgical technique, the preoperative and postoperative treatment will be identical for all subjects. Radiographic examinations of the feet (x-rays) will be made preoperatively and at two weeks postoperative and 12 weeks postoperative, as per the usual and customary practice of the principal investigator.

The conventional surgical technique is a Chevron-type distal metatarsal osteotomy, which is performed through a dorsomedial incision approximately 7 cm long. And osteotomy of the distal portion of the first metatarsal is made. The capital or distal fragment of the metatarsal is mobilized and displaced laterally an adequate amount to correct the hallux valgus deformity. The capital or distal fragment is stabilized in corrected position with screws. The internal fixation screws used in the conventional surgical technique do not require removal. Through the same incision, the contracted soft tissues on the lateral aspect of the metatarsophalangeal joint are released. Per the patient's request and consent, other planned bony or soft tissue pathology of the lesser toes that requires surgical correction (eg, hammer toes) will be treated in the same surgical session using standard techniques.

The minimally invasive surgical technique is a transverse subcapital distal metatarsal osteotomy, which is performed through a direct medial incision approximately 1 cm long. The osteotomy of the distal portion of the first metatarsal is made using fluoroscopic image guidance. The capital or distal fragment of the metatarsal is mobilized and displaced laterally an adequate amount to correct the hallux valgus deformity. A 2.0 mm Kirschner wire is placed percutaneously in a position medial to the proximal phalanx, and advanced proximally using fluoroscopic guidance until the proximal end of the wire is located in a stable position within the medullary cavity of the first metatarsal (see figures) .The distal end of the Kirschner wire is left outside the skin where it is cut to length and covered. The Kirschner wire is removed after six weeks. The soft tissues on the lateral aspect of the joint are not released. Per the patient's request and consent, other planned bony or soft tissue pathology of the lesser toes that requires surgical correction (e.g., hammer toes) will be treated in the same surgical session using standard techniques.

Postoperative Care -

* First post operative is: one week postoperative
* Second postoperative visit: two weeks postoperative
* Third postoperative visit: 6 weeks postoperative
* Last postoperative visit: 12 weeks postoperative

Period of Long Term Follow Up

* 1 year follow up - completion of questionnaire. This can be completed by email, regular mail, or in person, depending on the patients preference.
* 2 year follow up - completion of questionnaire. This can be completed by email, regular mail, or in person, depending on the patients preference.
* 3 year follow up - completion of questionnaire. This can be completed by email, regular mail, or in person, depending on the patients preference.

Study Costs

All costs associated with the usual and customary perioperative, operative, and postoperative care of the patients will be billed to the patient's medical insurance. Subjects will incur no costs that are solely for the purposes of research. Any study costs for the purposes of the research study will be supported by the principal investigator. These costs are not expected to be large. The main cost will be the time needed to inform the patient of the study process, obtain consent, gather the data and store it. The PI feels that unsupported research is a feasible and preferable alternative to industry funded studies, which have been shown to be much more likely to have significant bias.

Randomization and Blinding

After a study subject has been enrolled, they will be randomized to one of two treatment groups. All subjects will be randomized, 1:1 either to the conventional surgery group (group A) or the minimally invasive surgery (group B). Randomization will take place after enrollment via selection of a one of a multitude of envelopes containing a random number. A block randomization technique will be used with a block size of eight. Each random number will have been preassigned to either group A or group B.

The envelope containing the patient's group assignment will be opened in the operating room immediately prior to commencing the surgery. Due to the nature of the surgery, neither the investigators nor the patients can be effectively blinded to the results of the group assignment. The patients will be made aware of the group assignment after the surgery.

Primary outcomes measure and secondary outcomes measure

The primary outcomes measure is the Manchester-Oxford Foot Questionnaire Score (MOXFQ). Manchester-Oxford Foot Questionnaire' (MOXFQ), a 16 item patient-reported questionnaire.

Secondary outcome measures are preoperative to postoperative change in hallux valgus angle (HVA).

Data Collection and Statistical Analysis

The study documents will be labeled with the patients random number, and the data will be stored using only this unique random number identifier. The patient's name and group assignment will not appear on any study document. Data related to the MOXFQ will be recorded on a visit summary document bearing only the patient's random number, and later entered into a computerized spreadsheet using the patient's random number as a unique identifier. The patients personal data will not be stored along with the aggregate data. Data will be kept in a password secured computer in the office of the PI.

Power Analysis

Power analysis was performed using G*Power 3.0.10 (Department of Experimental Psychology Heinrich-Heine-University 40225 Düsseldorf Germany - http://www.psycho.uni-duesseldorf.de/aap/projects/gpower/). Power was calculated for the differences of two independent means (two groups). Given an estimated population effect size (d) of 0.65, a probability of alpha error (significance) of 0.05, and a required power (1- beta) of 0.80, the total required sample size would be 78 (two groups of 39). The two-tailed test is used because we cannot assume that the differences in the treatment effect in the two groups will be in one direction only, that is, we have assumed that the treatment effect may either be smaller or larger in the conventional surgery group than in the minimally invasive surgery group. Our goal is to enroll 80 patients in the trial. For independent samples, the Mann-Whitney test will be used to examine the difference between the two groups.

Study Endpoints

The study endpoint will occur when a sufficient number of patients have completed the 36 month long term follow-up process. Our aim is to enroll a minimum of 60 and a maximum of 100 patients. Once the last patient enrolled has completed the 36 month survey instrument, the data collection phase of the study will be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Patients with mild to moderate hallux valgus which has been unresponsive to nonoperative measures. Mild to moderate hallux valgus deformity is defined by weightbearing xray-findings of a hallux valgus angle of greater than normal (< 15°) and less than 39°, and a intermetatarsal angle less than 18°.
3. Patients who are willing to be randomized to either of the surgical procedures.
4. Patients who are able to understand and sign the consent form
5. Patients who are able to understand and complete the study questionnaires
6. Females with no documented evidence of current pregnancy, and willingness to take the necessary precautions to prevent pregnancy for the duration of the active participation period (12 weeks).

Exclusion Criteria:

1. Patients who have had previous bunion surgery on the affected foot
2. Patients who have symptomatic arthritis of the metatarsophalangeal joint (hallux rigidus).
3. History of systemic inflammatory condition or infection of the great toe or nearby soft tissues
4. Diabetic or neuropathic Charcot arthropathy
5. Significant vascular insufficiency
6. Factors which unacceptably increase the risk of surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Manchester-Oxford Foot Questionnaire Score (MOXFQ). | 12 months from date of surgery
  Manchester-Oxford Foot Questionnaire' (MOXFQ), a 16 item patient-reported questionnaire consisting of three domains/scales: 'Walking/standing' (seven items), 'Pain' (five items) and 'Social interaction' (four items). The MOXFQ is a validated disease-specific outcomes scale for foot and ankle surgery which has been shown to be responsive and reliable.

SECONDARY OUTCOMES:
2 weeks preoperative to 12 weeks postoperative change in hallux valgus angle (HVA). | 12 weeks
  Radiographic outcomes parameters will be measured using weight-bearing radiographs to analyze preoperative and postoperative hallux valgus angle, and the correction or normalization thereof. (Degrees of correction = preoperative HVA - 12 week postoperative HVA.)

CONTACTS AND LOCATIONS:
Locations (1):
- Newton Wellesley Hospital, Newton, Massachusetts, United States

REFERENCES:
- [Background] Smith SE, Landorf KB, Butterworth PA, Menz HB. Scarf versus chevron osteotomy for the correction of 1-2 intermetatarsal angle in hallux valgus: a systematic review and meta-analysis. J Foot Ankle Surg. 2012 Jul-Aug;51(4):437-44. doi: 10.1053/j.jfas.2012.02.016. Epub 2012 Apr 8. PMID 22487651
- [Background] Maffulli N, Longo UG, Marinozzi A, Denaro V. Hallux valgus: effectiveness and safety of minimally invasive surgery. A systematic review. Br Med Bull. 2011;97:149-67. doi: 10.1093/bmb/ldq027. Epub 2010 Aug 14. PMID 20710024
- [Background] Oliva F, Longo UG, Maffulli N. Minimally invasive hallux valgus correction. Orthop Clin North Am. 2009 Oct;40(4):525-30, x. doi: 10.1016/j.ocl.2009.06.005. PMID 19773058
- [Background] Ferrari J, Higgins JP, Prior TD. WITHDRAWN: Interventions for treating hallux valgus (abductovalgus) and bunions. Cochrane Database Syst Rev. 2009 Apr 15;2009(2):CD000964. doi: 10.1002/14651858.CD000964.pub3. PMID 19370560
- [Background] Deenik A, van Mameren H, de Visser E, de Waal Malefijt M, Draijer F, de Bie R. Equivalent correction in scarf and chevron osteotomy in moderate and severe hallux valgus: a randomized controlled trial. Foot Ankle Int. 2008 Dec;29(12):1209-15. doi: 10.3113/FAI.2008.1209. PMID 19138485